CLINICAL TRIAL: NCT04084054
Title: Ultrasonic Measurement of the Optic Nerve Sheath Diameter Predicting Outcome After Cardiac Arrest
Acronym: ONSD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NL71331.091.19
Record Dates: First submitted 2019-08-29; First posted 2019-09-10 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Post-Anoxic Coma
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasound — Ultrasonic measurement of the optic nerve sheath diameter

SUMMARY:
Rationale: An important proportion of patients with return of spontaneous circulation (ROSC) after cardiac arrest remain comatose as a result of post anoxic encephalopathy (PAE). Specific treatments to promote cerebral recovery are lacking. Early identification of patients without potential of recovery of brain functioning may prevent inappropriate continuation of medical treatment and improve communication between doctors and families. Intensivists currently use a combination of diagnostic measures, including brainstem reflexes, motor response, status myoclonus, SSEP measurements and (increasingly) the EEG. However, together all these measure identify only 20-50% of the patients with severe PAE precluding cerebral recovery. At the moment, there is a high demand for bedside measurements that contribute to the neurological prognostication of comatose patients after cardiac arrest. Non-invasive bedside measurements of the optic nerve sheath diameter (ONSD) using ultrasound hold potential to improve outcome prediction.

Objective: To estimate the value and feasibility of repetitive measurements of the ONSD in comatose patients after cardiac arrest.

Study design: Prospective cohort study

Study population: 160 subsequent comatose adult patients after cardiac arrest, admitted to the ICU of Rijnstate hospital

Intervention: In addition to standard treatments, patients will undergo ultrasonic measurements of the ONSD during the first 3 days after cardiac arrest. Survivors will be followed upon hospital discharge. ONSD measurements will be followed over time and related tot neurological outcome.

Main study parameters/endpoints: The primary outcome measure is neurological outcome, defined using the Cerebral Performance Category (CPC) score at 6 months. CPC 1-2 indicates favourable neurological outcome, and CPC 3-5 indicates unfavourable neurological outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Cardiac arrest
* Admitted to the ICU with Glasgow Coma Scale ≤ 8

Exclusion Criteria:

* Pregnancy
* Traumatic head injury
* Eye surgery in medical history, including cataract surgery
* Pre-existing dependency in daily living (CPC 3 or 4)
* Any known progressive brain illness, such as a brain tumour or neurodegenerative disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 160 subsequent comatose adult patients after cardiac arrest, admitted to the ICU of Rijnstate hospital.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2019-12-02 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Glasgow Coma Scale | At 6 months after cardiac arrest
  Neurological outcome, defined using the Cerebral Performance Category (CPC). CPC 1-2 indicates favourable neurological outcome, and CPC 3-5 indicates unfavourable neurological outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Rijnstate Hospital, Arnhem, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Robba C, Santori G, Czosnyka M, Corradi F, Bragazzi N, Padayachy L, Taccone FS, Citerio G. Optic nerve sheath diameter measured sonographically as non-invasive estimator of intracranial pressure: a systematic review and meta-analysis. Intensive Care Med. 2018 Aug;44(8):1284-1294. doi: 10.1007/s00134-018-5305-7. Epub 2018 Jul 17. PMID 30019201
- [Derived] Verhulst MMLH, Visser IM, Keijzer HM, de Kruijf NLM, Peters EJG, Wilbers T, Peelen RV, Hofmeijer J, Blans MJ. Additional predictive value of optic nerve sheath diameter for neurological prognosis after cardiac arrest: a prospective cohort study. Ultrasound J. 2023 Dec 8;15(1):46. doi: 10.1186/s13089-023-00344-3. PMID 38063930